CLINICAL TRIAL: NCT03801070
Title: Radiological Predictors of Failure of Endoscopic Therapy or Need For Multiple Endoscopic Procedures in Patients With Walled Off Pancreatic Necrosis
Brief Title: Rad Predictors for WON
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Oklahoma Medical Center (Unknown); Northwestern University Chicago Illinois (Unknown); St. Luke's Hospital, Kansas City, Missouri (Other)
Responsible Party: Sponsor
Other Study IDs: 201707053
Record Dates: First submitted 2019-01-03; First posted 2019-01-11 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Walled Off Pancreatic Necrosis (WON)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Less than median number necrosectomies: Group one includes patients who underwent less than median number necrosectomies
  Interventions: Procedure: endoscopic drainage of walled off pancreatic necrosis
- At least the median number of necrosectomies: Group two includes patients who underwent at least the median number of necrosectomies
  Interventions: Procedure: endoscopic drainage of walled off pancreatic necrosis

INTERVENTIONS:
Procedure: endoscopic drainage of walled off pancreatic necrosis — transmural drainage and mechanical debridement of solid debris (necrosectomy)

SUMMARY:
This is a retrospective chart review study examining 1) demographic data such as age, sex, etiology of pancreatitis 2) clinical data including radiological characteristics of walled off pancreatic necrosis, walled off necrosis related admissions and readmission following endoscopic drainage, surgical or percutaneous procedures performed for the management of walled off pancreatic necrosis, and clinical outcomes following treatment of WON (including hospital readmissions, WON resolution, procedure complications, WON related death) 3) endoscopy data including indication for initial endoscopic drainage and subsequent endoscopic procedures performed for management of walled off necrosis (including additional EGD's, endoscopic drainage procedures, and/or necrosectomy)

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who underwent endoscopic drainage of walled off pancreatic necrosis
* Patients who did not require further intervention (either surgical, percutaneous, or endoscopic) following endoscopic drainage
* Patients who required further intervention for walled off pancreatic necrosis (either surgical, percutaneous, or endoscopic) following endoscopic drainage.
* Patients who underwent percutaneous or surgical interventions prior to endoscopic drainage

Exclusion Criteria:

* Pancreatic pseudocysts without any solid debris
* Under 18 years of age at the time of endoscopic drainage

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with organized collections that contain both solid and liquid debris and arise from necrotizing pancreatitis, referred to as walled off pancreatic necrosis (WON)
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Identify WON imaging characteristics on cat-scan | through study completion, an average of 260 days
  Characteristics on cat-scan that are predictive of requiring multiple endoscopic procedures, percutaneous drainage, and/or surgical intervention for management of walled off pancreatic necrosis
Endoscopic course (total number and type of endoscopic treatments required for resolution of walled off necrosis, occurrence of treatment related complications) | through study completion, an average of 260 days
  Imaging classification method to efficiently report these imaging characteristics
Clinical course (number of hospital readmissions during treatment, rates of walled off necrosis resolution, rates of walled off necrosis related death) | through study completion, an average of 260 days
  Characteristics to develop a predictive model that will help to identify patients at high risk for requiring multiple endoscopic procedures, percutaneous drainage, and/or surgical intervention for management of walled off pancreatic necrosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine in St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No